CLINICAL TRIAL: NCT06156787
Title: Patterns of Urinary Bladder Cancer in Darfur, Sudan 2020 - 2022
Brief Title: Patterns of Urinary Bladder Cancer in Darfur, Suda
Status: Completed | Type: Observational
Sponsor: National Center for Gastroentestinal and Liver Disease (Other)
Responsible Party: Sponsor
Other Study IDs: ElbagieaBladder
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Background: Bladder cancer (BC) exhibits extreme heterogeneity regarding clinical outcome, etiology, histology, and geographic distribution. Recent clinical observations point to alterations in the BC pattern in the Sudan, possibly as a result of lifestyle changes brought on by the enormous migration from rural to urban locations. This study aimed to identify the pattern of bladder cancer in Darfur.

Patients and Methods: A cross sectional, hospital-based study, it was conducted inNyala specialized hospital, during the period from (2020 to 2022), included one hundred and five patients with bladder mass matching the inclusion criteria were studied over the diversity of demographic data , clinical finding, pathological type and possible risk factors .

ELIGIBILITY:
Inclusion Criteria:

* All Sudanese pts who lives in Darfur and presented with urinary bladder mass.
* Adult above 18 years

Exclusion Criteria:

* Patient who does not live in Darfur.
* Patients refused to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sudanese patients present to the urology department with urinary bladder mass
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Patterns of Urinary Bladder Cancer in Darfur, Sudan | The research is a cross-sectional, hospital-based study conducted at Nyala Specialized Hospital in Darfur. The study spans a period from 2020 to 2022.
  This research study investigates the patterns of urinary bladder cancer (BC) in Darfur, Sudan, with a focus on understanding the clinical outcomes, etiology, histology, and demographic distribution of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Nyala specialized hospital, Darfur, Darfur, Sudan